CLINICAL TRIAL: NCT04055090
Title: Long-term, Prospective, Non-interventional, Extension of a Phase III, Randomized, Placebo-controlled, Multicenter Study to Assess the Safety & Efficacy of Engensis (VM202) in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Extension of Phase 3 Gene Therapy for Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMDN-003b
Record Dates: First submitted 2019-02-22; First posted 2019-08-13 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Painful Diabetic Neuropathy; Diabetic Neuropathy, Painful
Keywords: diabetic; neuropathy; shooting pain; burning pain; pins and needles pain; foot pain; ViroMed; Helixmith; Engensis; VM202
MeSH Terms: conditions — Diabetic Neuropathies; Pain

STUDY DESIGN:
Intervention Model Description: Long term, prospective, non-interventional, safety extension study of phase 3 trial. Double blind, randomized, placebo-controlled, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects who received Engensis (VM202) (Experimental): VM202, Engensis
  Interventions: Genetic: Long-Term Follow-Up of Patients who Received Engensis (VM202)
- Subjects who received Placebo (Placebo Comparator): Placebo, vehicle
  Interventions: Drug: Long-Term Follow-Up of Patients who Received Placebo

INTERVENTIONS:
Genetic: Long-Term Follow-Up of Patients who Received Engensis (VM202) — No study drug is administered in this study. Patients who received Engensis (VM202) in the previous trial (VMDN-003) will remain blinded and were evaluated in this trial for long-term safety and efficacy.
  Arms: Subjects who received Engensis (VM202)
Drug: Long-Term Follow-Up of Patients who Received Placebo — No study drug is administered in this study. Patients who received Placebo in the previous trial (VMDN-003) will remain blinded and were evaluated in this trial for long-term safety and efficacy.
  Arms: Subjects who received Placebo

SUMMARY:
The purpose of this study is to explore the overall safety profile and durability of efficacy of Engensis (VM202) in painful diabetic peripheral neuropathy.

All subjects still in follow-up for the VMDN-003 study or who have completed the Day 270 visit within the prior 90 days will be approached to enroll in the long-term safety extension study.

DETAILED DESCRIPTION:
In the phase III VMDN-003 study, subjects received 2 treatments of either Engensis (VM202) or placebo administered as intramuscular injections into bilateral calves on Days 0 and 14, and Days 90 and 104. Primary efficacy was evaluated 90 days following the first injection. The growth potential for Hepatocyte Growth Factor make long-term follow-up important both for safety and efficacy: in order for Engensis to be a candidate for chronic treatment of Painful Diabetic Peripheral Neuropathy, it must be demonstrated not to induce unexpected adverse events with repeated dosing; and the potential for reversal or stabilization of diabetic neuropathy using only one or two treatments of Engensis may make it especially attractive compared to current treatments which must be taken daily for the duration of the disease. A safety extension to the VMDN-003 study is therefore warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Were randomized and dosed in the VMDN-003 study
2. Received all intramuscular injections of study drug on Days 0, 14, 90, and 104 in the VMDN-003 study
3. Were in follow-up for the VMDN-003 study or had completed Day 270 within the last 90 days prior to signing consent

Exclusion Criteria:

1. Were using an investigational drug or treatment
2. Were unable or unwilling to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Kessler, MD, Principal Investigator — Northwestern University
Locations (14):
- United States (14):
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Northern California Research, Sacramento, California
  - Center for Clinical Research, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of West Florida, Clearwater, Florida
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Nerve and Muscle Center of Texas, Houston, Texas
  - EVMS (Eastern Virginia Medical School), Norfolk, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Who Received Engensis (VM202): VM202- Engensis
  Long-Term Follow-Up of Patients who Received Engensis (VM202): No study drug is administered in this study.
  Patients who received Engensis (VM202) in a previous trial will be evaluated in this trial for long-term safety and efficacy.
- Subjects Who Received Placebo: Placebo, vehicle
  Long-Term Follow-Up of Patients who Received Placebo: No study drug is administered in this study.
  Patients who received Placebo in a previous trial will be evaluated in this trial for long-term safety and efficacy.
Period: Overall Study
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Started (Treatment assignments (Engensis or Placebo) for this study, VMDN-003b, are based on the treatment groups in the prior study, VMDN-003) | 65 | 36
Completed | 63 | 36
Not Completed | 2 | 0
Not completed — screen failure | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who signed consent for the safety extension study. Participants in the safety analysis population were analyzed according to the treatment received in the VMDN-003 study, regardless of the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo | Total
Number analyzed (Participants) | 65 | 36 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 20 | 52
  >=65 years | 33 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.87) | 61.4 (8.98) | 61.5 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 8 | 33
  Male | 40 | 28 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 1 | 1 | 2
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 9 | 5 | 14
  Race: White | 53 | 28 | 81
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 65 | 36 | 101
Gabapentin and/or Pregabalin Use [Count of Participants; unit: Participants] | 31 | 17 | 48
Diabetes Type [Count of Participants; unit: Participants] — Population: The race for one subject who screen failed was missing
  Participants
    Type I diabetes | 2 | 2 | 4
    Type II diabetes | 62 | 34 | 96
    Not reported | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (4.79) | 33.2 (5.45) | 32.9 (5.01)
HbA1c [Mean (Standard Deviation); unit: percent of glycosylated hemoglobin] | 7.37 (1.19) | 7.22 (0.95) | 7.31 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety for Engensis Versus Placebo
Description: Long-term (6 months) safety in terms of the incidence of Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events for Subjects who received Engensis or Placebo (in the prior VMDN-003 study)
Time Frame: Baseline through Day 365
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Who Received Engensis (VM202): VM202- Engensis
  Long-Term Follow-Up of Patients who Received Engensis (VM202): No study drug is administered in this study.
  Patients who received Engensis (VM202) in the previous trial (VMDN-003) will remain blinded and were evaluated in this blinded trial for long-term safety and efficacy.
- Subjects Who Received Placebo: Placebo, vehicle
  Long-Term Follow-Up of Patients who Received Placebo: No study drug is administered in this study.
  Patients who received placebo in the previous trial (VMDN-003) will remain blinded and were evaluated in this blinded trial for long-term safety and efficacy.
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Number analyzed (Participants) | 65 | 36
Participants
  Subjects with at least one Treatment-emergent Adverse Event (TEAE) | 10 | 8
  Subjects with at least one Treatment-emergent Serious Adverse Event (TESAE) | 1 | 2

2. Secondary Outcome: The Change in the Average 24-hour Pain Score From Baseline (Day 0 of Study VMDN-003) to Day 365 for Engensis Versus Placebo
Description: The Average 24-hour Pain Score was obtained from the Daily Pain and Sleep Interference Diary. The change in the Average 24-hour Pain Score was determined from baseline (Day 0 of Study VMDN-003) to the Day 365 visit. The Average 24-hour Pain Score is an 11-point numerical scale with scores from 0 (No Pain) to 10 (Worst Possible Pain).
Time Frame: Baseline to the Day 365
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Subjects Who Received Engensis (VM202): VM202- Engensis
  Long-Term Follow-Up of Patients who Received Engensis (VM202): No study drug is administered in this study.
  Patients who received Engensis (VM202) in the previous trial (VMDN-003) will remain blinded and were evaluated in this trial for long-term safety and efficacy.
- Subjects Who Received Placebo: Placebo, vehicle
  Long-Term Follow-Up of Patients who Received Placebo: No study drug is administered in this study.
  Patients who received Placebo in the previous trial (VMDN-003) will remain blinded and were evaluated in this trial for long-term safety and efficacy.
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Number analyzed (Participants) | 65 | 36
score on a scale | -2.32 (2.36) | -1.49 (1.76)
Statistical Analysis 1: Comparison: Subjects Who Received Engensis (VM202) vs Subjects Who Received Placebo; Test type: Other; p = 0.0460, Mixed Models Analysis; Mixed-effects Model for Repeated Measures (MMRM) with treatment, visit, treatment-by-visit, and use of gabapentin/pregabalin as main fixed effects; Least Square Mean Difference = -0.89, 95% CI 2-sided [-1.76 to -0.02], Standard Error of Mean 0.438 — Mixed-effects Model for Repeated Measures with treatment, visit, treatment-by-visit, and use of gabapentin/pregabalin as main fixed effects. The Baseline average 24-hour pain score was included as a covariate

3. Secondary Outcome: Change in the Average 24-hour Pain Score From Day 270 to Day 365 for Engensis Versus Placebo
Description: The Average 24-hour Pain Score is from the Daily Pain and Sleep Interference Diary. The change in the Average 24-hour Pain Score was determined for Day 270 to Day 365. The Average 24-hour Pain Score is an 11-point numerical scale with scores from 0 (No Pain) to 10 (Worst Possible Pain).
Time Frame: Day 270 to Day 365
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Number analyzed (Participants) | 65 | 36
score on a scale | 0.26 (1.525) | 0.29 (1.430)

4. Secondary Outcome: Patient's Global Impression of Change at the Day 365 Visit for Engensis Versus Placebo
Description: The Patient's Global Impression of Change was completed by subjects (self-administered) at the Day 365 visit. The subject evaluated how his/her overall status had changed since the start of the study using a 7-point Patient's Global Impression of Change questionnaire scale, where 1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, and 7 = Very Much Worse.
  The Outcome Measure was the Patient's Global Impression of Change Categories of Scores as follows: 1 = Very Much Improved or Much Improved, 0 = Minimally Improved/Worsened or No Change, and -1 = Much Worse or Very Much Worse.
Time Frame: At the Day 365 visit
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Number analyzed (Participants) | 65 | 36
Participants
  1: Very much improved or much improved | 31 | 14
  0: Minimally improved/worsened or no change | 31 | 20
  -1: Much worse or very much worse | 1 | 2
  Not Reported | 2 | 0
Statistical Analysis 1: Comparison: Subjects Who Received Engensis (VM202) vs Subjects Who Received Placebo; Test type: Other; p = 0.2190, Cochran-Mantel-Haenszel

5. Secondary Outcome: Subgroup Analysis of the Change in the Average 24-hour Pain Score From Baseline (Day 0 of Study VMDN-003) to Day 365 for Engensis Versus Placebo for Subjects Without Gabapentin and/or Pregabalin Use at Baseline
Description: The Average 24-hour Pain Score was obtained from the Daily Pain and Sleep Interference Diary and the change in the Average 24-hour Pain Score from baseline (Day 0 of Study VMDN-003) to the Day 365 follow-up was determined. The Average 24-hour Pain Score is an 11-point numerical scale with scores from 0 (No Pain) to 10 (Worst Possible Pain).
Time Frame: Baseline to Day 365
Population: Intent-to-Treat population subgroup analysis of Subjects without gabapentin and/or pregabalin use
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
Number analyzed (Participants) | 34 | 19
score on a scale | -2.30 (0.352) | -0.82 (0.470)
Statistical Analysis 1: Comparison: Subjects Who Received Engensis (VM202) vs Subjects Who Received Placebo; Test type: Other; p = 0.0155, Mixed Models Analysis; Least-Squares Mean Difference = -1.48, 95% CI 2-sided [-2.67 to -0.29] — Mixed-effects Model for Repeated Measures (MMRM) with treatment, visit, treatment-by-visit, and use of gabapentin/pregabalin as main fixed effects. Baseline average 24-hour pain score is included as a covariate

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 270 (start of VMDN-003b study) to Day 365
Description: Treatment-emergent adverse events
Arm/Group | Subjects Who Received Engensis (VM202) | Subjects Who Received Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/65 | 2/36
Other Adverse Events (participants affected / at risk) | 10/65 | 8/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Who Received Engensis (VM202) (N=65) | Subjects Who Received Placebo (N=36)
acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Who Received Engensis (VM202) (N=65) | Subjects Who Received Placebo (N=36)
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator Agreement

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04055090/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04055090/SAP_001.pdf